CLINICAL TRIAL: NCT06684990
Title: Evaluation of a Fast Point-of-care Platform for Diabetes Care at Out-patient Clinics
Brief Title: Point-of-Care Testing in Outpatient Diabetes Care
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Taichung Veterans General Hospital (Other)
Responsible Party: Principal Investigator, Jun-Sing Wang, MD, PhD, Director, Division of Endocrinology and Metabolism, Taichung Veterans General Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: CE24395C
Record Dates: First submitted 2024-11-08; First posted 2024-11-12 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Diabetes
Keywords: Diabetes; HbA1c; cystatin C; point of care
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: The investigators will conduct POC testing for HbA1c and cystain C in outpatients with diabetes, and present the results to their providers. Follow up data on fasting glucose, HbA1c, serum creatinine, urine albumin to creatinine ratio (UACR), lipids profile, ...etc will be collected every 6 months for 3 years. Patients who decline to POC testing but provide consent to observational follow up will serve as the controls. The investigators will examine the effects of POC testing on changes in glycemic control and renal function in study participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Outpatients with diabetes who provide consent to POC testing (Experimental): Intervention: POC testing for HbA1c and cystatin C. Observational follow up: data on fasting glucose, HbA1c, serum creatinine, urine albumin to creatinine ratio (UACR), lipids profile, ...etc.
  Interventions: Other: POC testing
- Outpatients with diabetes who decline to POC testing, but consent to observational follow up (No Intervention): This group will serve as the controls. Follow up data on fasting glucose, HbA1c, serum creatinine, urine albumin to creatinine ratio (UACR), lipids profile, ...etc.

INTERVENTIONS:
Other: POC testing — POC testing for HbA1c and cystatin C
  Arms: Outpatients with diabetes who provide consent to POC testing

SUMMARY:
Using a point-of-care (POC) platform, the investigators will investigate the effects of POC testing for glycated hemoglobin (HbA1c) and cystatin C at out-patient clinics on long-term diabetes outcomes.

DETAILED DESCRIPTION:
Laboratory testing for HbA1c and cystatin C is time-consuming, and healthcare providers often do not have update results when they evaluate outpatients with diabetes. A POC testing platform may help address this issue, and the investigators aim to examine its effects on diabetes outcomes.

ELIGIBILITY:
Inclusion Criteria:

-Adults aged 18 to 80 receiving treatment and follow-up for diabetes at outpatient clinics of Taichung Veterans General Hospital, Taichung, Taiwan.

Exclusion Criteria:

1. Past medical history of hemolytic anemia, hemoglobinopathies (sickle cell anemia HbS, fetal hemoglobin HbF), iron deficiency anemia, thalassemia, pernicious anemia, recent blood transfusions, acute bleeding requiring erythropoiesis-stimulating agents.
2. Chronic liver disease, cirrhosis, hyperbilirubinemia, asplenia (splenomegaly, splenectomy).
3. Hypertriglyceridemia (over 500 mg/dl), or alcoholism.
4. Thyroid dysfunction, active malignant tumors under treatment, HIV infection.
5. Long-term use (over three months) of steroids or cyclosporine.
6. Severe proteinuria (e.g., nephrotic syndrome), or a baseline eGFR <60 ml/min/1.73 m².

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 222 (Actual)
Dates: Start 2025-01-02 (Actual); Primary Completion 2028-04 (Estimated); Study Completion 2028-04 (Estimated)

PRIMARY OUTCOMES:
Changes from baseline to the end of study in eGFR | Observational follow up period of 3 years
  Estimated glomerular filtration rate (eGFR) will be determined using the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) equation (Levey AS, et al. Ann Intern Med. 2009; 150: 604-12).

SECONDARY OUTCOMES:
Changes from baseline to the end of study in UACR | Observational follow up period of 3 years

OTHER OUTCOMES:
Incident chronic kidney disease | Observational follow up period of 3 years
  incident chronic kidney disease is defined as an eGFR <60 ml/min/1.73 m2 of at least 3 months duration.

CONTACTS AND LOCATIONS:
Locations (1):
- Taichung Veterans General Hospital, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided
Data will be available from the principal investigator on reasonable request.